CLINICAL TRIAL: NCT04151108
Title: The Copenhagen PROTECT Study: Biomarkers for Length of Hospital Stay and Loss of Muscle Mass and Function in Old Medical Patients
Brief Title: Biomarkers for Length of Hospital Stay and Loss of Muscle Mass and Function in Old Medical Patients
Acronym: PROTECT
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Charlotte Suetta, Professor, MD, Dr.Med., Bispebjerg Hospital
Other Study IDs: H-19039214
Record Dates: First submitted 2019-10-28; First posted 2019-11-05 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Sarcopenia; Muscle Loss; Length of Stay
MeSH Terms: conditions — Sarcopenia; Muscular Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — Plasma and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Old medical patients: Blood tests, frailty (CSHA Frailty Scale), risk of pressure ulcers (Braden Score), handgrip strength, chair-rise test, Orientation-Memory-Concentration test (OMC), screening for sarcopenia (SARC-F), screening for malnutrition (SNAQ), body composition.
  Will be assessed at admission
  Interventions: Other: Development of a risk assessment tool based on clinical and functional measures and systemic biomarkers
- Geriatric patients: Blood tests, frailty (CSHA Frailty Scale), risk of pressure ulcers (Braden Score), handgrip strength, chair-rise test, gait-speed, Orientation-Memory-Concentration test (OMC), screening for sarcopenia (SARC-F), screening for malnutrition (SNAQ), body composition.
  Blood tests, physical function measures and body composition will be assessed at both admission and discharge.
  Interventions: Other: Development of a risk assessment tool based on clinical and functional measures and systemic biomarkers; Other: Development of a risk assessment tool for loss of muscle mass and physical function based on clinical and functional measures and systemic biomarkers

INTERVENTIONS:
Other: Development of a risk assessment tool based on clinical and functional measures and systemic biomarkers — Blood tests, frailty (CSHA Clinical Frailty Scale) and risk of pressure ulcers (Braden Score), Early Warning Score (EWS), sarcopenia (SARC-F), malnutrition (SNAQ), cognitive status, comorbidity (Charlson comorbidity Index), polypharmacy, muscle strength, and body composition (BIA)
Other: Development of a risk assessment tool for loss of muscle mass and physical function based on clinical and functional measures and systemic biomarkers — Blood tests, frailty (CSHA Clinical Frailty Scale), Early Warning Score (EWS), cognitive status, sarcopenia (SARC-f), malnutrition (SNAQ), comorbidity (Charlson comorbidity Index), polypharmacy, physical function, physical performance, and body composition (BIA)
  Groups: Geriatric patients

SUMMARY:
As humans age, there is a gradual loss of skeletal muscle mass and strength, termed sarcopenia. The underlying causes of sarcopenia are yet not fully elucidated but are thought to be multifactorial and include increased levels of systemic pro-inflammatory mediators, a decrease in anabolic hormones and changes in the neuromuscular system. Furthermore, physical inactivity, chronic diseases, immobilisation and hospitalisation are known to play an important part in the development of sarcopenia.

The prevalence of sarcopenia ranges from 20-30% (aged >70yrs) within the general community. However, the prevalence of sarcopenia in geriatric patients after an acute hospital admission is substantially higher, estimated at ≈50%. Furthermore, successive events of hospitalisation have been suggested to contribute to the development of sarcopenia, as even short periods (4-5 days) of skeletal muscle disuse are known to induce muscle atrophy.

Mean length of hospital stay in geriatric wards due to acute illness or hip-fracture is typically 7 to 11 days during which the level of physical activity is strongly reduced leading to an accelerated loss of muscle mass that many older patients never recover from.

Notably, a substantial part of the deterioration in functional capacity could be avoided just by counteracting loss of muscle mass during hospitalization. As such, we need to identify sensitive biological, clinical and functional biomarkers predicting loss of muscle mass and function during hospitalization to identify patients at risk of developing sarcopenia. Additionally, it is crucial to investigate the association of these biomarkers with hospital length of stay, as hospitalisation has been suggested to contribute to the development of sarcopenia while longer hospital stays may increase patient risk of hospital-acquired infections and place an economic burden on society.

ELIGIBILITY:
Inclusion Criteria:

* equal to or over the age of 65
* admitted to the acute ward at Bispebjerg Hospital

Exclusion Criteria:

* age under 65 years
* terminal illness
* participants who do not understand Danish
* participants in isolation with airborne or droplet infections

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will consist of participants admitted to the acute ward and the geriatric ward at Bispebjerg Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1072 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Length of stay | From date of hospital admission until discharge, assessed up to 2 months
  Hours of admission from index to discharge
Change in muscle mass | Change from baseline muscle mass, assessed at admission, to muscle mass assessed at discharge, an average of 10 days
  Relative change in muscle mass during hospitalization
Change in muscle strength | Change from baseline muscle strength, assessed at admission, to muscle strength assessed at discharge, an average of 10 days
  Change in handgrip strength during hospitalization
Change in physical function | Change from baseline physical function, assessed at admission, to physical function assessed at discharge, an average of 10 days
  Change in chair-rise and gait-speed ability during hospitalization

SECONDARY OUTCOMES:
Readmission | Time to readmission 90 days from discharge
  Time to readmission from discharge
Mortality | Time to mortality 90 days from index admission
  Time to mortality from index admission

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Suetta, Professor, Principal Investigator — Geriatric Research Unit, Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
The following will be available: Study Protocol and Statistical Analysis Plan (SAP).

REFERENCES:
- [Derived] Kamper RS, Schultz M, Hansen SK, Andersen H, Ekmann A, Nygaard H, Helland F, Wejse MR, Rahbek CB, Noerst T, Pressel E, Nielsen FE, Suetta C. Biomarkers for length of hospital stay, changes in muscle mass, strength and physical function in older medical patients: protocol for the Copenhagen PROTECT study-a prospective cohort study. BMJ Open. 2020 Dec 29;10(12):e042786. doi: 10.1136/bmjopen-2020-042786. PMID 33376179

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/08/NCT04151108/Prot_SAP_000.pdf